CLINICAL TRIAL: NCT01266161
Title: A Multiple Dose Dental Pain Study Of An Ibuprofen 600 Mg Extended Release Caplet
Brief Title: Multiple Dose Dental Pain Study Of Ibuprofen Extended Release
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B3491001; AK-10-13 (Other: Alias Study Number)
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Pain
Keywords: dental pain; multiple dose; ibuprofen; third molar extraction
MeSH Terms: conditions — Pain; Toothache | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibuprofen 600 mg extended release (Experimental)
  Interventions: Drug: Ibuprofen 600 mg ER
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen 600 mg ER — One 600 mg caplet dosed at 0, 12, 24 and 36 hours
  Arms: Ibuprofen 600 mg extended release
Drug: Placebo — One placebo caplet dosed at times 0, 12, 24 and 36 hours
  Arms: Placebo

SUMMARY:
The study hypothesis is that single and multiple doses of ibuprofen 600 mg ER caplets provide analgesic efficacy superior to placebo over 12-hour dosing intervals.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16 to 40 years of age
* Subjects who undergo surgical removal of at least two third molars
* One of which must be a partial or full bony mandibular impaction
* Subjects must have at least moderate baseline pain (a score of 2 on the categorical pain severity rating scale) confirmed by a score of at least 50 mm on the 100-mm visual analog scale-pain severity rating scale (VAS-PSR)

Exclusion Criteria:

* Acute localized dental infection at the time of surgery that could confound the post-surgical evaluation
* Presence or history of any significant organ disease
* Use of prescription or OTC first generation antihistamines
* Females who are pregnant, lactating or of childbearing potential and not using a medically approved method to prevent pregnancy

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2010-11-22 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2011-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Central Texas Oral Surgery Associates, Austin, Texas
  - Premier Research, Austin, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3491001&StudyName=Multiple%20Dose%20Dental%20Pain%20Study%20Of%20Ibuprofen%20Extended%20Release

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo 1 matching caplet administered orally up to 5 hours after surgery, thereafter every 12 hours up to 48 hours
- Ibuprofen: Ibuprofen 600 milligrams (mg) extended release (ER) caplet administered orally up to 5 hours after surgery, thereafter every 12 hours up to 48 hours
Period: Overall Study
Arm/Group | Placebo | Ibuprofen
Started | 52 | 54
Completed | 48 | 53
Not Completed | 4 | 1
Not completed — Ineligible | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Vomited within 4 hours of dosing | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen | Total
Number analyzed (Participants) | 52 | 54 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.1 (3.3) | 21.3 (3.6) | 21.2 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 19 | 18 | 37
Pain Severity [Number; unit: participants] — A 4-point categorical pain severity rating scale was used to rate the severity of baseline pain in response to the query " My starting pain is:" Responses ranged and were scored as follows: None (0), Mild (1), Moderate (2), Severe (3). A baseline pain intensity score of at least moderate was required for study enrollment.
  participants
    Moderate | 37 | 39 | 76
    Severe | 15 | 15 | 30
Pain Intensity [Mean (Standard Deviation); unit: millimeter] — A 100-millimeter (mm) visual analog scale-pain severity rating (VAS-PSR) rated intensity of baseline pain. Participants were asked to "Draw a single vertical line on the scale that shows how much pain you have at this time." Scores on this 100-mm linear scale measured to nearest millimeter from left. Zero on the scale represented no pain and 100 represented the worst pain. Score of at least 50 mm required for enrolment.
  millimeter | 73.8 (12.25) | 75.7 (12.18) | 74.8 (12.20)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of Pain Relief and Pain Intensity Difference Scores From 0 to 12 Hours After the First Dose (SPRID 0-12)
Description: SPRID is time-weighted sum of pain relief (PR) plus pain intensity (PI) difference (PID) (PRID) scores. 5-point categorical scale for PR: "How much relief do you have from your starting pain?" (0 equals [=] none, 1=a little, 2=some, 3=a lot, 4=complete). 4-point categorical scale for PI: "How much pain do you have at this time?" (0=none, 1=mild, 2=moderate, 3=severe). PID score=baseline pain intensity score minus pain intensity at each time point; score ranged from -1 to 3; higher positive PID value indicated improvement in pain intensity. SPRID 0-12 score ranged from -12 to 84; higher score indicated better efficacy.
Time Frame: Baseline to 12 hours
Population: Intent-to-treat (ITT) population: Randomized participants with at least moderate baseline pain (score 2 on the pain severity rating [PSR] scale) confirmed by a score of at least 50 millimeter (mm) on the 100-mm visual analog scale (VAS)-PSR, within approximately 5 hours after surgery, provided a baseline assessment, and received study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale | 18.2 (20.0) | 41.5 (21.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Test type: Superiority; p < 0.001, ANOVA — p-Value from analysis of variance (ANOVA) model, with treatment, baseline PSR, gender terms. To protect type I error at 5% significance, 2 primary parameters tested sequentially: SPRID 8-12 not declared significant unless SPRID 0-12 was significant; Mean Difference (Final Values) = 23.76, 95% CI 2-sided [16.45 to 31.07]

2. Primary Outcome: Sum of Pain Relief and Pain Intensity Difference Scores From 8-12 Hours After the First Dose
Description: SPRID is time-weighted sum of PR plus PID (PRID) scores. 5-point categorical scale for PR: "How much relief do you have from your starting pain?" (0=none, 1=a little, 2=some, 3=a lot, 4=complete). 4-point categorical scale for pain intensity: "How much pain do you have at this time?" (0=none, 1=mild, 2=moderate, 3=severe). PID score=baseline pain intensity score minus pain intensity at each time point; score ranged from -1 to 3; higher positive PID value indicated improvement (decrease) in pain intensity. SPRID 8-12 score ranged from -4 to 28; higher score indicated better efficacy.
Time Frame: 8 to 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale | 10.3 (12.0) | 18.4 (12.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model, with treatment, baseline PSR, and gender terms. To protect type I error at 5% significance, 2 primary parameters tested sequentially: SPRID 8-12 not declared significant unless SPRID 0-12 was significant; Mean Difference (Final Values) = 8.42, 95% CI 2-sided [4.13 to 12.71]

3. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference (SPID) Scores
Description: SPID is a derived endpoint from PID scores. For pain intensity, "How much pain do you have at this time?" answered on a 4-point categorical scale (0=none, 1=mild, 2=moderate, 3=severe). PID score=baseline pain intensity score minus pain intensity at each time point; score ranged from -1 to 3; higher positive PID value indicated improvement (decrease) in pain intensity. SPID scores ranged as follows: 0 to 12 hour (-11.5 to 35.5), 8 to 12 hour (-6.0 to 18.0), 12 to 24 hour (-14.0 to 42.0), 20 to 24 hour (-8.0 to 24.0), 0 to 24 hour (-23.5 to 71.5), 24 to 36 hour (-16.0 to 48.0), 32 to 36 hour (-8.0 to 24.0), 36 to 48 hour (-16.0 to 48.0), 44 to 48 hour (-8.0 to 24.0), 24 to 48 hour (-28.0 to 84.0); higher positive values indicated improvement (decrease) in pain intensity.
Time Frame: 0 to 12 hours, 8 to 12 hours, 12 to 24 hours, 20 to 24 hours, 0 to 24 hours, 24 to 36 hours, 32 to 36 hours, 36 to 48 hours, 44 to 48 hours, 24 to 48 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  SPID 0-12 | 4.1 (9.6) | 12.8 (9.5)
  SPID 8-12 | 2.5 (5.4) | 5.5 (5.2)
  SPID 12-24 | 12.5 (12.5) | 18.7 (11.7)
  SPID 20-24 | 8.8 (7.5) | 10.7 (7.3)
  SPID 0-24 | 15.5 (19.3) | 29.9 (18.8)
  SPID 24-36 | 16.2 (15.2) | 21.6 (13.9)
  SPID 32-36 | 7.0 (7.8) | 10.2 (7.4)
  SPID 36-48 | 17.4 (14.2) | 23.0 (13.8)
  SPID 44-48 | 10.5 (7.7) | 12.7 (7.3)
  SPID 24-48 | 30.5 (25.2) | 40.7 (23.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; For SPID 0-12; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 8.95, 95% CI 2-sided [5.94 to 11.95]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; For SPID 8-12; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 3.15, 95% CI 2-sided [1.45 to 4.85]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; For SPID 12-24; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 6.56, 95% CI 2-sided [2.84 to 10.27]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen; For SPID 20-24; Test type: Superiority; p = 0.091, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 2.02, 95% CI 2-sided [-0.33 to 4.37]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; For SPID 0-24; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 14.95, 95% CI 2-sided [9.12 to 20.79]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen; For SPID 24-36; Test type: Superiority; p = 0.010, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 5.87, 95% CI 2-sided [1.42 to 10.33]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen; For SPID 32-36; Test type: Superiority; p = 0.004, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 3.48, 95% CI 2-sided [1.13 to 5.83]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen; For SPID 36-48; Test type: Superiority; p = 0.006, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 6.09, 95% CI 2-sided [1.82 to 10.36]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen; For SPID 44-48; Test type: Superiority; p = 0.042, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 2.41, 95% CI 2-sided [0.09 to 4.73]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen; For SPID 24-48; Test type: Superiority; p = 0.004, ANOVA — p-Value from ANOVA model with treatment, baseline PSR, and gender terms; Least-squares means = 10.97, 95% CI 2-sided [3.49 to 18.45]

4. Secondary Outcome: Time to First Dose of Rescue Medication After First Dose of Study Drug
Description: During the first 12 hours of the study, participants not experiencing adequate relief after the 1-hour time point were allowed to take a single tablet (dose) of acetaminophen/hydrocodone hydrochloride (HCl) 500 mg/5 mg as a rescue medication (the only rescue medication allowed). The time at which rescue medication was taken was recorded.
Time Frame: Baseline to 12 hours
Population: ITT population. Here, "Number of participants analysed signifies those participants who were evaluable for this outcome measures".
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 40 | 16
hours | 1.6 [1.4 to 2.2] | NA [NA to NA] — Median time was more than 12 hours. 95% CI was not estimable.
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Test type: Superiority; p < 0.001, proportional hazards model; Hazard Ratio (HR) = 0.18, 95% CI [0.10 to 0.34]

5. Secondary Outcome: Percentage of Participants Taking Rescue Medication
Description: Participants not experiencing adequate relief after the 1-hour time point during each dosing interval were allowed to take a single tablet (dose) of acetaminophen/hydrocodone HCl 500 mg/5 mg as a rescue medication (the only rescue medication allowed) during each interval.
Time Frame: Baseline to 48 hours
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
percentage of participants
  First dosing interval (0 to 12 hours) | 76.9 | 29.6
  Second dosing interval (12 to 24 hours) | 30.8 | 5.6
  Third dosing interval (24 to 36 hours) | 32.7 | 9.3
  Fourth dosing interval (36 to 48 hours) | 19.2 | 5.6
  Overall during the study (0 to 48 hours) | 78.8 | 31.5
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; During the first dosing interval (0 to 12 hours); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Values from the Cochran-Mantel-Haenszel (CMH) test, controlling for baseline PSR and gender; Treatment Difference = -48.01, 95% CI [-64.46 to -31.56]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; During the second dosing interval (12 to 24 hours); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Values from the CMH test, controlling for baseline PSR and gender; Treatment Difference = -25.53, 95% CI [-39.78 to -11.28]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; During the third dosing interval (24 to 36 hours); Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — p-Values from the CMH test, controlling for baseline PSR and gender; Treatment Difference = -24.05, 95% CI [-38.93 to -9.18]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen; During the fourth dosing interval (36 to 48 hours); Test type: Superiority; p = 0.035, Cochran-Mantel-Haenszel — p-Values from the CMH test, controlling for baseline PSR and gender; Treatment Difference = -13.60, 95% CI [-26.41 to -0.79]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; During the study overall (0 to 48 hours); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Values from the CMH test, controlling for baseline PSR and gender; Treatment Difference = -48.01, 95% CI [-64.42 to -31.60]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen; Time to First Dose Rescue Medication Over Entire Study Period (0-48 Hours); Test type: Superiority; p = 0.011, Andersen-Gill (AG); Cox proportional hazard models = 0.086, 95% CI 2-sided [0.01 to 0.57]

6. Secondary Outcome: Pain Relief (PR) Scores
Description: A 5-point categorical pain relief rating scale was used to rate pain relief in response to the question: "How much relief do you have from your starting pain?" Responses were scored as follows: 0=none, 1=a little, 2=some, 3=a lot, 4=complete. Higher score indicated more pain relief.
Time Frame: 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  0.5 hours | 0.4 (0.7) | 1.3 (1.1)
  1 hour | 0.7 (1.0) | 2.2 (1.2)
  1.5 hours | 0.6 (1.0) | 2.6 (1.3)
  2 hours | 0.5 (1.0) | 2.8 (1.2)
  4 hours | 0.7 (1.3) | 2.9 (1.3)
  6 hours | 1.9 (1.3) | 2.8 (1.1)
  8 hours | 1.4 (1.3) | 2.4 (1.3)
  10 hours | 1.0 (1.3) | 2.1 (1.4)
  12 hours | 1.5 (1.5) | 1.9 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 0.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.84, 95% CI [0.50 to 1.19]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1 hour; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.53, 95% CI [1.11 to 1.94]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 2.00, 95% CI [1.56 to 2.44]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 2 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 2.29, 95% CI [1.86 to 2.73]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 4 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 2.18, 95% CI [1.69 to 2.68]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 6 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.92, 95% CI [0.46 to 1.38] — Treatment difference (ibuprofen minus placebo) and corresponding 95% CI were calculated based on least-squares means from the ANOVA model
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 8 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.04, 95% CI [0.54 to 1.54]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 10 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.10, 95% CI [0.59 to 1.60]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 12 hours; Test type: Superiority; p = 0.052, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.50, 95% CI [-0.00 to 1.01]

7. Secondary Outcome: Pain Intensity Difference (PID) Scores
Description: For pain intensity, "How much pain do you have at this time?" answered on a 4-point categorical scale. Responses were scored as follows: 0=none, 1=mild, 2=moderate, 3=severe. PID score=baseline pain intensity score minus score at each time point. PID scores ranged from -1 to 3. Higher positive PID scores indicated greater improvement (decrease in pain intensity).
Time Frame: 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  0.5 hours | 0.1 (0.6) | 0.5 (0.7)
  1 hour | 0.1 (0.8) | 1.0 (0.9)
  1.5 hours | 0.0 (0.9) | 1.2 (0.9)
  2 hours | -0.0 (0.8) | 1.4 (1.0)
  4 hours | 0.1 (1.0) | 1.4 (1.0)
  6 hours | 0.7 (1.0) | 1.3 (0.9)
  8 hours | 0.4 (0.9) | 1.0 (1.0)
  10 hours | 0.3 (0.9) | 0.9 (0.9)
  12 hours | 0.5 (1.2) | 0.8 (0.9)
  16 hours | 0.7 (0.9) | 1.6 (0.9)
  20 hours | 1.0 (1.0) | 1.4 (0.9)
  24 hours | 1.2 (1.0) | 1.2 (0.9)
  28 hours | 1.1 (1.1) | 1.6 (1.0)
  32 hours | 1.0 (1.0) | 1.6 (1.0)
  36 hours | 0.8 (1.0) | 1.0 (1.0)
  40 hours | 0.9 (1.0) | 1.6 (0.9)
  44 hours | 1.3 (1.0) | 1.6 (0.9)
  48 hours | 1.4 (1.0) | 1.6 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 0.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.37, 95% CI [0.16 to 0.59]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1 hour; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 0.90, 95% CI [0.63 to 1.18]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 1.22, 95% CI [0.91 to 1.52]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 2 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 1.40, 95% CI [1.10 to 1.71]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 4 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 1.32, 95% CI [0.97 to 1.67]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 6 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 0.61, 95% CI [0.30 to 0.91]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 8 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 0.64, 95% CI [0.31 to 0.97]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 10 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 0.66, 95% CI [0.36 to 0.97]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 12 hours; Test type: Superiority; p = 0.089, ANOVA — p-Values from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 0.27, 95% CI [-0.04 to 0.59]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 16 hours; Test type: Superiority; p < 0.001, ANOVA — Ibuprofen versus placebo at 0.5 hours; Least squares means = 1.00, 95% CI [0.70 to 1.29]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 20 hours; Test type: Superiority; p = 0.004, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.47, 95% CI [0.15 to 0.78]
Statistical Analysis 12: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 24 hours; Test type: Superiority; p = 0.821, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.04, 95% CI [-0.28 to 0.35]
Statistical Analysis 13: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 28 hours; Test type: Superiority; p = 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.56, 95% CI [0.23 to 0.90]
Statistical Analysis 14: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 32 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.62, 95% CI [0.30 to 0.94]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 36 hours; Test type: Superiority; p = 0.127, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.25, 95% CI [-0.07 to 0.57]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 40 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.67, 95% CI [0.35 to 1.00]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 44 hours; Test type: Superiority; p = 0.036, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.34, 95% CI [0.02 to 0.67]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 48 hours; Test type: Superiority; p = 0.091, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.26, 95% CI [-0.04 to 0.56]

8. Secondary Outcome: Pain Relief Combined With Pain Intensity (PRID) Scores
Description: PRID score=PR plus PID. 5-point categorical scale for PR: "How much relief do you have from your starting pain?" (0=none, 1=a little, 2=some, 3=a lot, 4=complete). 4-point categorical scale for pain intensity: "How much pain do you have at this time?" (0=none, 1=mild, 2=moderate, 3=severe). PID score=baseline pain intensity score minus pain intensity at each time point; PID score ranged from -1 to 3; higher positive PID value=improvement. PRID scores ranged from -1 to 7. Higher PRID scores indicated better pain relief and decrease in pain intensity.
Time Frame: 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  0.5 hours | 0.6 (1.1) | 1.8 (1.6)
  1 hour | 0.8 (1.7) | 3.2 (2.0)
  1.5 hours | 0.6 (1.7) | 3.8 (2.2)
  2 hours | 0.5 (1.7) | 4.1 (2.1)
  4 hours | 0.8 (2.2) | 4.3 (2.2)
  6 hours | 2.5 (2.2) | 4.0 (1.9)
  8 hours | 1.8 (2.1) | 3.5 (2.2)
  10 hours | 1.3 (2.0) | 3.0 (2.2)
  12 hours | 2.0 (2.6) | 2.7 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 0.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.22, 95% CI [0.69 to 1.74]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1 hour; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 2.43, 95% CI [1.77 to 3.09]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 1.5 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 3.22, 95% CI [2.49 to 3.95]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 2 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 3.70, 95% CI [2.98 to 4.42]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 4 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 3.50, 95% CI [2.67 to 4.33]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 6 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.53, 95% CI [0.79 to 2.27]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 8 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.67, 95% CI [0.87 to 2.48]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 10 hours; Test type: Superiority; p < 0.001, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 1.76, 95% CI [0.97 to 2.54]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 12 hours; Test type: Superiority; p = 0.056, ANOVA — p-Values from ANOVA model with treatment, baseline PSR, and gender terms; Least squares means = 0.78, 95% CI [-0.02 to 1.58]

9. Secondary Outcome: Time-weighted Sum of Pain Relief Scores (TOTPAR)
Description: TOTPAR is a derived endpoint from PR scores. 5-point categorical scale for PR: "How much relief do you have from your starting pain?" (0=none, 1=a little, 2=some, 3=a lot, 4=complete). TOTPAR 0-12 scores ranged from 0 (worst) to 48 (best). TOTPAR 8-12 scores ranged from 0 (worst) to 16 (best).
Time Frame: 0-12 hours, 8-12 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  TOTPAR 0 to 12 | 14.1 (11.2) | 28.7 (12.3)
  TOTPAR 8 to 12 | 7.8 (7.2) | 12.9 (7.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 0 to 12 hours; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 14.82, 95% CI 2-sided [10.38 to 19.25]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo from 8 to 12 hours; Test type: Superiority; p < 0.001, ANOVA — p-Value from ANOVA model with treatment, baseline pain severity, and gender terms; Least squares means = 5.27, 95% CI 2-sided [2.57 to 7.98]

10. Secondary Outcome: Number of Doses of Rescue Medication Used
Time Frame: 0-12, 12-24, 24-36, 36-48, 0-48 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
doses
  First dosing interval (0-12 hours) | 1.3 (1.0) | 0.4 (0.6)
  Second dosing interval (12-24 hours) | 0.4 (0.6) | 0.1 (0.2)
  Third dosing interval (24-36 hours) | 0.5 (0.9) | 0.1 (0.5)
  Fourth dosing interval (36-48 hours) | 0.3 (0.7) | 0.1 (0.3)
  Overall during the study (0-48 hours) | 2.5 (2.6) | 0.6 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; For the first dosing interval; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Values from the CMH test with modified ridit scores, controlling for baseline PSR and gender; CMH-adjusted proportion = -0.73, 95% CI 2-sided [-0.91 to -0.55]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; For the second dosing interval; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Treatment difference (ibuprofen minus placebo) and corresponding 95% CI were calculated based on CMH-adjusted proportions and corresponding standard errors; CMH-adjusted proportions = -0.72, 95% CI 2-sided [-1.05 to -0.40]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen; For the third dosing interval; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel — p-Values from the CMH test with modified ridit scores, controlling for baseline PSR and gender; CMH-adjusted proportions = -0.48, 95% CI 2-sided [-0.90 to -0.06]
Statistical Analysis 4: Comparison: Placebo; For the fourth dosing interval; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel — p-Values from the CMH test with modified ridit scores, controlling for baseline PSR and gender; CMH-adjusted proportion = -0.68, 95% CI 2-sided [-1.02 to -0.35]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen; For the overall study duration; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Values from the CMH test with modified ridit scores, controlling for baseline PSR and gender; CMH-adjusted proportion = -0.70, 95% CI 2-sided [-0.89 to -0.51]

11. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: The elapsed time from dosing until the participant indicated first perceptible pain relief by pressing the first stopwatch, provided the participant also indicated achieving meaningful relief by pressing the second stopwatch. Perceptible relief defined as when participant first began to feel any pain-relieving effect whatsoever of the drug. Did not necessarily mean the participant felt completely better, but when the participant first felt any difference in the pain he/she is currently feeling.
Time Frame: Baseline to 12 hours
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 17 | 48
minutes | NA [NA to NA] — Median time to first perceptible relief was more than 720 minutes. 95% CI was not estimable. | 25.0 [20.1 to 28.5]

12. Secondary Outcome: Time to Meaningful Relief
Description: Participants evaluated the time to meaningful relief by depressing a second stopwatch at the moment they first began to experience meaningful relief, defined as relief from the pain that was considered meaningful to the participant.
Time Frame: Baseline to 12 hours
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 17 | 48
minutes | NA [NA to NA] — Time to meaningful relief was more than 720 minutes. 95% CI not calculated. | 54.2 [46.5 to 79.6]

13. Secondary Outcome: Participant Global Evaluation Score
Description: Participants responded, on a 6-point categorical scale, to the following question: "How would you rate this medication as a pain-reliever?" Responses on this categorical scale ranged as follows: 0=very poor, 1=poor, 2=fair, 3=good, 4=very good, 5=excellent.
Time Frame: 24 and 48 hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen
Number analyzed (Participants) | 52 | 54
units on a scale
  24 hours | 1.2 (1.4) | 3.5 (1.2)
  48 hours | 1.7 (1.5) | 3.7 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 24 hours; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — p-Value from the CMH test with modified ridit scores, controlling for baseline PSR score and gender; Gamma statistic = 0.85, 95% CI 2-sided [0.74 to 0.95]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen; Ibuprofen versus placebo at 48 hours; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; p-Value from the CMH test with modified ridit scores, controlling for baseline PSR score and gender; Gamma statistic = 0.79, 95% CI 2-sided [0.66 to 0.92]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/54
Other Adverse Events (participants affected / at risk) | 23/52 | 8/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Ibuprofen (N=54)
Ear pain (Ear and labyrinth disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 1
Vomiting (Gastrointestinal disorders) | 6 | 0
Chills (General disorders) | 1 | 0
Feeling hot (General disorders) | 2 | 0
Flushing (General disorders) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 9 | 4
Skin burning sensation (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.